CLINICAL TRIAL: NCT00806260
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Cross-over Study to Evaluate the Psychomotor Effect of VI-0521 in Healthy Overweight and Obese Subjects.
Brief Title: A Study to Evaluate How VI-0521 Affect Psychomotor Performance in Healthy Overweight and Obese Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: MDS Pharma Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OB-205
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-08

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; coordination; psychomotor
MeSH Terms: conditions — Overweight; Obesity | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment 1 (Experimental): Dosed first with alcohol, then active VI-0521, and last, VI-0521 placebo
  Interventions: Drug: VI-0521; Drug: Placebo; Other: Alcohol
- Treatment 2 (Experimental): First dosed with alcohol placebo (fruit juice), then active VI-0521, and last, placebo VI-0521
  Interventions: Drug: VI-0521; Drug: Placebo; Other: alcohol placebo
- Treatment 3 (Experimental): First dosed with alcohol, then VI-0521 placebo, and last, active VI-0521
  Interventions: Drug: VI-0521; Drug: Placebo; Other: Alcohol
- Treatment 4 (Experimental): First dosed with alcohol placebo, then VI-0521 placebo, and last, active VI-0521
  Interventions: Drug: VI-0521; Drug: Placebo; Other: alcohol placebo

INTERVENTIONS:
Drug: VI-0521 — Phentermine 3.75 mg and topiramate 23 mg daily for the 1st week; Phentermine 7.5 mg and topiramate 46 mg daily for the 2nd week; Phentermine 11.25 mg and topiramate 69 mg daily for the 3rd week; Phentermine 15 mg and topiramate 92 mg daily for the 4th week
Drug: Placebo — Placebo daily for 4 weeks
Other: Alcohol
  Arms: Treatment 1; Treatment 3
Other: alcohol placebo — fruit juice
  Arms: Treatment 2; Treatment 4

SUMMARY:
The purpose of this study is to determine how VI-0521 affect speed and reaction time on specific tasks that require eye and hand coordination, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Written consents;
* Adequate contraception from screening through 28 days after the last dose of study drug for female subjects;
* Healthy obese or overweight subjects with BMI between 27 and 35.

Exclusion Criteria:

* History of glaucoma or any past or present use of medications to treat increased intraocular pressure;
* Current use of any tobacco products, including cigarettes, cigars, pipes, or chewing tobacco, or use within the three months prior to screening;
* History of drug abuse during the three years prior to screening;
* History of alcohol abuse, or excessive alcohol consumption, or describes themselves as non-users of alcohol;
* Current depression of moderate or greater severity, or any presence or history of suicidal behavior or active suicidal ideation
* More than one lifetime episode of major depression;
* Currently working night shifts at a job;
* On average consumes greater than two cups of coffee or xanthine-containing beverages per day (>200 mg/day) within the two weeks prior to screening;
* Any use of dietary, herbal, and/or fitness/body-building supplements (with the exception of vitamins) within one month prior to screening;
* Aspartate aminotransferase or alanine aminotransferase >2.5 x ULN;
* Serum creatinine ≥1.5 mg/dL for men or ≥1.4 mg/dL for women.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Peterson, Study Director — VIVUS LLC; Alan Marion, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- Research Site, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred within the US between January 2009 and March 2009
Pre-assignment Details: Period 1 was not a crossover design. Subjects were randomized to either alcohol or alcohol-placebo. Subjects who completed Period 1 were then randomized to the crossover portion of the study, Periods 2 and 3.
Groups:
- Alcohol, VI-0521 Placebo Then VI-0521: Alcohol was administered during period one followed by one week washout, VI-0521 placebo for four weeks during period two followed by one week washout, then VI-0521 titrated over four weeks during period three.
- Alcohol, VI-0521 Then VI-0521 Placebo: Alcohol was administered during period one followed by one week washout, VI-0521 titrated over four weeks during period two followed by one week washout, then VI-0521 placebo for four weeks during period three.
- Alcohol-placebo, VI-0521-placebo Then VI-0521: Alcohol-placebo was administered during period one followed by one week washout, VI-0521 placebo for four weeks during period two followed by one week washout, then VI-0521 titrated over four weeks during period three.
- Alcohol-placebo, VI-0521 Then VI-0521-placebo: Alcohol-placebo was administered during period one followed by one week washout, VI-0521 titrated over four weeks during period two followed by one week washout, then VI-0521 placebo for four weeks during period three.
- Alcohol Only: Alcohol was administered during period one after which the subject's participation ended.
- Alcohol-placebo Only: Alcohol-placebo was administered during period one after which the subject's participation ended.
Period: Period 1 (1 Day)
Arm/Group | Alcohol, VI-0521 Placebo Then VI-0521 | Alcohol, VI-0521 Then VI-0521 Placebo | Alcohol-placebo, VI-0521-placebo Then VI-0521 | Alcohol-placebo, VI-0521 Then VI-0521-placebo | Alcohol Only | Alcohol-placebo Only
Started | 15 | 8 | 8 | 14 | 18 | 17
Completed | 15 | 8 | 8 | 14 | 15 (did not move onto Periods 2 and 3 due to adjusted design of study) | 17 (did not move onto Periods 2 and 3 due to adjusted design of study)
Not Completed | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3 | 0
Period: Period 2
Arm/Group | Alcohol, VI-0521 Placebo Then VI-0521 | Alcohol, VI-0521 Then VI-0521 Placebo | Alcohol-placebo, VI-0521-placebo Then VI-0521 | Alcohol-placebo, VI-0521 Then VI-0521-placebo | Alcohol Only | Alcohol-placebo Only
Started | 15 | 8 | 8 | 14 | 0 | 0
Completed | 13 | 8 | 6 | 12 | 0 | 0
Not Completed | 2 | 0 | 2 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Need to take concomitant medication | 1 | 0 | 0 | 0 | 0 | 0
Not completed — sponsor request | 0 | 0 | 1 | 1 | 0 | 0
Period: Period 3
Arm/Group | Alcohol, VI-0521 Placebo Then VI-0521 | Alcohol, VI-0521 Then VI-0521 Placebo | Alcohol-placebo, VI-0521-placebo Then VI-0521 | Alcohol-placebo, VI-0521 Then VI-0521-placebo | Alcohol Only | Alcohol-placebo Only
Started | 13 | 8 | 6 | 12 | 0 | 0
Completed | 12 | 7 | 5 | 12 | 0 | 0
Not Completed | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alcohol, VI-0521 Placebo Then VI-0521: Participants in this study arm were given alcohol in period 1, VI-0521 placebo in period 2 and VI-0521 in period 3.
- Alcohol, VI-0521 Then VI-0521 Placebo: Participants in this study arm were given alcohol in period 1, VI-0521 in period 2 and VI-0521-placebo in period 3.
- Alcohol Placebo, VI-0521 Placebo Then VI-0521: Participants in this study arm were given alcohol placebo in period 1, VI-0521-placebo in period 2 and VI-0521 in period 3.
- Alcohol Placebo, VI-0521 Then VI-0521 Placebo: Participants in this study arm were given alcohol placebo in period 1, VI-0521 in period 2 and VI-0521 placebo in period 3.
- Alcohol Only: Subjects in this study arm only participated in period 1 and were given alcohol.
- Alcohol Placebo Only: Subject in this study arm only participated in period 1 and were given alcohol placebo.
- Total: Total of all reporting groups
Arm/Group | Alcohol, VI-0521 Placebo Then VI-0521 | Alcohol, VI-0521 Then VI-0521 Placebo | Alcohol Placebo, VI-0521 Placebo Then VI-0521 | Alcohol Placebo, VI-0521 Then VI-0521 Placebo | Alcohol Only | Alcohol Placebo Only | Total
Number analyzed (Participants) | 15 | 8 | 8 | 14 | 18 | 17 | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 26.7 (5.4) | 29.9 (7.8) | 31.1 (8.6) | 27.4 (6.1) | 30.1 (7.7) | 27.4 (6.3) | 28.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 1 | 6 | 7 | 1 | 21
  Male | 10 | 7 | 7 | 8 | 11 | 16 | 59
Region of Enrollment [Number; unit: participants]
  United States | 15 | 8 | 8 | 14 | 18 | 17 | 80

OUTCOME MEASURES:

1. Primary Outcome: Measure of Psychomotor Function Using Speed and Coordination on the CogScreen Pathfinder Number (PFN) Test in Subjects Treated With Alcohol Compared to Alcohol Placebo in Period 1.
Description: CogScreen-Psychomotor Edition (CogScreen-PM) consists of a series of computerized cognitive tasks, each self-contained and presented with instructions and a practice segment. The test battery takes about 20-25 minutes to perform. Performance on the test will be measured as the median reaction time for correct responses (PFNRTC) and coordination errors (PFNCOOR) before and after treatment. The measures of the tests are:
  (a) response speed, the median response time to complete each sequential step (PFNRTC); (b) response accuracy (PF Number Accuracy [PFNACC]); and (c) a coordination measure indicating the respondent's proximity to the center of the target numbers and letters (PF Number Coordination [PFNCOOR]). PF measures number sequencing skills, immediate memory, psychomotor speed and coordination, and visual scanning.
  The normal range for PFN scores is 1.17-2.16. Scores that are higher than this range indicate some level of psychomotor impairment.
Time Frame: at breath alcohol levels 0.10%, 0.07%, and 0.04%
Population: modified-intent-to-treat (mITT)
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Period 1 Alcohol-placebo: fruit juice
- Period 1 Alcohol: Alcohol
Arm/Group | Period 1 Alcohol-placebo | Period 1 Alcohol
Number analyzed (Participants) | 23 | 23
scores on a scale
  Breath Alcohol Level 0.10% | 1.57 (0.06) | 1.90 (0.06)
  Breath Alcohol Level 0.07% | 1.67 (0.04) | 1.88 (0.05)
  Breath Alcohol Level 0.04% | 1.62 (0.05) | 1.68 (0.05)
Statistical Analysis 1: Comparison: Period 1 Alcohol-placebo vs Period 1 Alcohol; at alcohol level 0.10%; Test type: Non-Inferiority or Equivalence — step down test; ANCOVA; Mean Difference (Final Values) = 0.33, 90% CI 1-sided [lower limit 0.21], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Period 1 Alcohol-placebo vs Period 1 Alcohol; at alcohol level 0.07%; Test type: Non-Inferiority or Equivalence — step down test; ANCOVA; Mean Difference (Final Values) = 0.21, 90% CI 1-sided [lower limit 0.12], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Period 1 Alcohol-placebo vs Period 1 Alcohol; at alcohol level 0.04%; Test type: Non-Inferiority or Equivalence — step-down test; ANCOVA; Mean Difference (Final Values) = 0.06, 90% CI 1-sided [lower limit -0.03], Standard Error of Mean 0.06

2. Primary Outcome: Measure of Psychomotor Function Using Speed and Coordination on the CogScreen Pathfinder Number (PFN) Test in Subjects Treated With VI-0521 Compared to Placebo in Periods 2 and 3.
Description: as for outcome 1
Time Frame: Hour 2 and Hour 6
Population: Intent-to-treat (ITT) ITT population includes participants who completed Periods 1, 2 and 3. Subjects that were discontinued due to adverse events, failed drug/alcohol screens, non-compliance, etc. are not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Period 2 VI-0521-placebo; Period 3 VI-0521-placebo: Placebo
- Period 2 VI-0521; Period 3 VI-0521: phentermine/topiramate
Arm/Group | Period 2 VI-0521-placebo | Period 2 VI-0521 | Period 3 VI-0521-placebo | Period 3 VI-0521
Number analyzed (Participants) | 36 | 36 | 36 | 36
scores on a scale
  Hour 2 | 1.69 (0.04) | 1.64 (0.04) | 1.65 (0.04) | 1.64 (0.04)
  Hour 6 | 1.67 (0.04) | 1.60 (0.04) | 1.65 (0.03) | 1.60 (0.03)
Statistical Analysis 1: Comparison: Period 2 VI-0521-placebo vs Period 2 VI-0521; at 2 hr timepoint; Test type: Non-Inferiority or Equivalence — non-inferiority; ANCOVA; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.17 to 0.07], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Period 2 VI-0521-placebo vs Period 2 VI-0521; at 6 hr timepoint; Test type: Non-Inferiority or Equivalence — non inferiority test; ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.18 to 0.04], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Period 3 VI-0521-placebo vs Period 3 VI-0521; at 2 hr timepoint; Test type: Non-Inferiority or Equivalence — non inferiority; ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.08 to 0.06], Standard Error of Mean 0.03
Statistical Analysis 4: Comparison: Period 3 VI-0521-placebo vs Period 3 VI-0521; at 6 hr timepoint; Test type: Non-Inferiority or Equivalence — non inferiority; ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.13 to 0.05], Standard Error of Mean 0.04

ADVERSE EVENTS:
Time Frame: AEs were collected from when written informed consent was provided through 28 days after the last dose of investigational product.
Groups:
- Period 2 and 3 Placebo: Total number of subjects that were given VI-0521 placebo was 43. 1 subject was excluded from the analysis due to failing a drug/alcohol screen leaving 42 subjects in the ITT population.
- Period 2 and 3 Qnexa: The total number of subjects that were given VI-0521 was 41. 2 subjects were excluded from the analysis, one due to failing a drug/alcohol screen and the other due to pregnancy. Excluding these two subjects leaves 39 subjects in the analyzed ITT population.
Arm/Group | Period 1 Placebo | Period 1 Alcohol | Period 2 and 3 Placebo | Period 2 and 3 Qnexa
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41 | 0/42 | 0/39
Other Adverse Events (participants affected / at risk) | 5/39 | 22/41 | 11/42 | 14/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 Placebo (N=39) | Period 1 Alcohol (N=41) | Period 2 and 3 Placebo (N=42) | Period 2 and 3 Qnexa (N=39)
diarrhea (Gastrointestinal disorders) | 2 | 2 | 1 | 1
dry mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 4
nausea (Gastrointestinal disorders) | 2 | 8 | 0 | 0
dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
pain (General disorders) | 0 | 2 | 0 | 2
disturbance in attention (Nervous system disorders) | 2 | 0 | 0 | 2
headache (Nervous system disorders) | 3 | 11 | 0 | 4
parethesia (Nervous system disorders) | 0 | 0 | 2 | 4
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2
hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Due to technical issues, an additional cohort of subjects were added to Period 1 only, which produced two additional treatment arms, alcohol only and alcohol placebo only. No change was made in the data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.